CLINICAL TRIAL: NCT05087108
Title: A Crossover Study of the Hemodynamic Effect of the OsciPulse Device Compared to Reference Therapies
Brief Title: Evaluation of the OsciPulse Rapid Cycling Compression Device Effects on Venous Blood Flow
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: OsciFlex LLC (Industry)
Collaborators: University of Pennsylvania (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OSC-VTE-002; R44HL145860 (NIH)
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-03

CONDITIONS: Venous Thromboses; Venous Stasis
Keywords: Venous compression; Intermittent pneumatic compression
MeSH Terms: conditions — Venous Thrombosis; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study arm (Experimental): In this single arm study all enrolled subjects will the intervention by the investigational device, and both reference devices. Ultrasound will be used to measure the blood flow in the subject during the use of all three devices.
  Interventions: Device: OsciPulse system; Device: Reference Therapy 1; Device: Refence Therapy 2

INTERVENTIONS:
Device: OsciPulse system — The OsciPulse system is an intermittent pneumatic limb compression system. The OsciPulse sleeves that are applied to the top portion of the user's calves and are periodically inflated with rapid bursts of compressed air to create frequent pulses of venous return.
Device: Reference Therapy 1 — The Venaflow Elite is a sequential compression device that uses compressed air to inflate sleeves worn on the calf of the user to stimulate venous return. The Venaflow system sleeves cover the entire calf region of the user and contain two bladders that are inflated sequentially to induce venous return.
  Other Names: Venaflow Elite Vascular System
Device: Refence Therapy 2 — The Kendall SCD device is a sequential compression device that uses compressed air to inflate sleeves worn on the calf of the user to stimulate venous return. The Kendall SCD sleeves cover the entire calf region of the user and contain three bladders that are inflated sequentially to induce venous return.
  Other Names: Kendall 700 Series SCD

SUMMARY:
This study will evaluate the effects on venous blood flow of the investigational device, OsciPulse system, which is an external intermittent limb compression device. The study will enroll healthy human subjects who will have their deep venous blood flow measured by vascular ultrasound during immobility, use of the OsciPulse system, and use of two reference vascular compression devices. Our hypothesis is that the OsciPulse system will create distinct patterns of venous flow, specifically at the site of venous valves, in comparison to the reference compression devices.

DETAILED DESCRIPTION:
Enrolled healthy subjects will undergo and initial vascular ultrasound imaging procedure to locate a deep venous valve in either the sapheno-femoral junction or femoral trifurcation sites. Once the imaging valve is identified the baseline level of venous flow will be collected in 30 s video clips of 2D color Doppler videos and spectral Doppler. Next, either the OsciPulse device, or one of the two reference therapy devices, will be applied by study personnel according to the device's specific instructions. The subject will wear the device during the capture of 1 spectral Doppler clip and three 30 s 2D color Doppler ultrasound clips on both the left and right leg. Next, the remaining two devices will be applied based on instructions, and vascular ultrasound clips captured for each. Completion of this visit protocol will be the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult age ≥40 years old
* Generally healthy.
* No history of diagnosed vascular disease including: DVT, PE, VTE, peripheral vascular disease, post-phlebitic syndrome, or chronic venous insufficiency.
* Mentally alert and understand English proficiently.
* Able to give informed consent.

Exclusion Criteria:

* Skin breaks, abrasion, or irritation in the area of the limb in contact with the OsciPulse device or reference therapies.
* Severe peripheral artery or venous disease.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Venous valve sinus forward flow volume index | Visit 1 - 60 minutes
  The volume flow index (mL/mL) will be measured for flow in the valve sinus region that is moving back towards the heart (forward flow). The venous flow at a valve will be measured using 2D color Doppler ultrasound, and flow volume index calculated from the resulting video clips.
Venous valve sinus reversing flow volume index | Visit 1 - 60 minutes
  The volume flow index (mL/mL) will be measured for flow in the valve sinus region that is moving away from the heart (reversing flow). The venous flow at a valve will be measured using 2D color Doppler ultrasound, and flow volume index calculated from the resulting video clips.
Deep vein centerline flow | Visit 1 - 60 minutes
  The velocity of venous flow measured by spectral Doppler ultrasound in the deep femoral vein.
Venous valve sinus rouleaux | Visit 1 - 60 minutes
  The degree of red blood cell rouleaux in the sinus of venous valves will be measured using B-mode ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: John Welsh, PhD, Study Director — OsciFlex LLC; Chandra Sehgal, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Our plan is to make available for sharing all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available starting 6 months after publication of the study and will be available for 24 months upon request.
Access Criteria: Qualifying IPD will be shared with specific requestors if they are at an academic or government institution and to be used for non-commercial research. Requests will be evaluated by OsciFlex LLC.